CLINICAL TRIAL: NCT06615830
Title: HIPANC-002 - Observational Performance Study of Transcriptome-Based OncoTreat/OncoTarget Testing With Patient-Derived Organoids in Metastatic Pancreatic Cancer
Brief Title: Predictive Value of Transcriptome-based OncoTreat/Oncotarget and Organoid Testing in Metastatic Pancreatic Cancer.
Status: Not yet recruiting | Type: Observational
Sponsor: Prof. Dr. med. Dres. h.c. Jan Schmidt, MME (Other)
Collaborators: Klinik Hirslanden, Zurich (Other); Insel Gruppe AG, University Hospital Bern (Other); Columbia Research Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Dres. h.c. Jan Schmidt, MME, Prof. Dr. med. Dres. h.c. MME, Klinik Hirslanden, Zurich
Organization: Klinik Hirslanden, Zurich (Other)
Other Study IDs: HIPANC_002
Record Dates: First submitted 2024-09-01; First posted 2024-09-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pancreas Neoplasms; Pancreatic Neoplasms; Pancreatic Cancer Metastatic; Pancreatic Adenocarcinoma Metastatic
Keywords: Pancreatic cancer; Pancreatic adenocarcinoma; Metastatic pancreatic adenocarcinoma; Organoid; Organoid-driven chemotherapy; Darwin Oncotreat; Darwin Oncotarget; Personalized chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pancreatic cancer tissue from metastasis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Predictive value of Oncotreat/Oncotarget testing in palliative chemotherapy in pancreatic cancer: The study will include patients with diagnosis of metastatic pancreatic adenocarcinoma. After complete disease staging, patients will undergo laparoscopic surgical biopsy of metastatic tumoral tissue. The tissue will serve for the generation of Oncotreat and Oncotarget tests as well as for patient-derived organoids on which potentially predicted drugs will be benchmarked.
  Each patient will receive the standard first-line and second-line chemotherapy (chosen among Gemcitabine-Abraxane, or Abraxane-Gemcitabine-FOLFOX or FOLFIRINOX, based on the clinical judgement of the treating oncologist).
  When progression occurs predictive value of the test with regard to Progression-free Survival (PFS) will be analyzed.

SUMMARY:
Pancreatic cancer is burdened by a survival of barely 10% at 5 years. About 80% of new cases do not qualify for surgery due to either locally-advanced or metastatic disease. In patients with good performance status (PS), palliative first-line treatments mainly consist of combination regimens, such as FOLFIRINOX, modified FOLFIRINOX or Gemcitabine-Abraxane. For subjects with a poor PS, instead, guidelines recommend single-agent infusions (e.g. Gemcitabine, Capecitabine or 5-FU alone). Nevertheless, upon disease progression therapeutic options are still scarce and with limited sustained efficacy.

Overall survival in metastatic pancreatic cancer ranges between 9.1 and 13.5 months, while progression-free survival under either FOLFIRINOX or Gemcitabine-Abraxane spans between 5.5 and 6.4 months. This timespan reduces even further when standard second-line regimens must be initiated upon disease progression.

Nowadays, genomic and transcriptomic analysis are crucial tools in cancer research that enable the identification of genetic mutations and alterations that drive the development and progression of cancer. By studying the changes in the DNA and RNA sequences of cancer cells, researchers can gain insights into the underlying molecular mechanisms of cancer and identify potential therapeutic targets. Genomic analysis can identify specific mutations or alterations that are present in cancer cells, while transcriptomic analysis can reveal changes in gene expression that may be linked to disease progression or response to treatment. These analyses are an essential component for the development of precision medicine approaches, which aim to tailor cancer treatment to the individual genetic profile of each patient.

PDOs can replicate in vitro the biological, genetic and molecular aspects of the primary tumour. Some of their advantages include their rapid growth compared to xenografts, the possibility to perform high-throughput drug screening, and their direct application to precision oncology by predicting best therapies. In this study they will be used as an in vitro comparator of the molecular tests to the clinical course of the patient.

Overall, combining genomic and transcriptomic analysis with PDO technology in cancer research might lead to exponential capacity to provide oncologic patients with extremely tailored and effective cancer treatments in the future.

For HIPANC-002 these tests are being evaluated as non-interventional investigational IVD's. Test results are not to be used for protocol mandated therapy decisions.

DETAILED DESCRIPTION:
Primary objective.

The study seeks primarily to demonstrate whether a significant correlation between the IVD based predicted drug sensitivity and the patient's progression-free survival (PFS) in metastatic pancreatic adenocarcinoma after administered standard therapies (which are not chosen based on the test) exist.

Secondary objectives. The study seeks further to

1. Explore the correlation between Darwin-test predicted drug sensitivity and patient-derived PDO sensitivity to clinically used drug regimens.
2. Explore the correlation between the measured PDO sensitivity to the administered standard therapies and the clinical course of the patient, i.e. PFS (in vivo and in vitro comparison).
3. Collect samples for biobanking and future identification of potential new markers associated with tumor response.

Safety objectives.

The study aims to assess:

The rate and severity of 30-days post-operative surgical complications related to laparoscopic surgical biopsy required to retrieve tumoral tissue for IVD-based testing and PDO generation.

The primary outcome is achieved if a significant correlation between IVD based predictions of drug sensitivity and clinically observed patient outcome (progression-free survival after administered standard therapy) exist.

The secondary outcomes are achieved if

1. There is a significant correlation between Darwin-test predicted drug sensitivity and patient-derived PDO sensitivity to clinically used drug regimens.
2. There is a significant correlation between the measured PDO sensitivity to the administered standard therapies and the clinical course of the patient, i.e. PFS (in vivo and in vitro comparison).

Biobanked samples will be retrospectively analysed to highlight potential biochemical markers of tumour response to therapy if attributable.

The safety outcome will assess descriptively the rate of severe surgical post-operative complication related to laparoscopic surgical biopsy required to retrieve tumoral tissue for IVD-testing and PDO generation and occurring within 30 postoperative days.

Non-Interventional, single arm, observational study

Inclusion criteria:

* Informed Consent as documented by signature
* Patients older than 18 years
* Patients with metastatic pancreatic ductal adenocarcinoma
* At least one lesion amenable for surgical excisional biopsy
* ECOG Performance status 0-2
* Radiologically measurable disease
* Life expectancy > 3 months
* Absolute leucocyte count >1.5 G/l, platelets >100 G/l
* Serum creatinine <1.5 times of the upper limit of normal or Clearance >50ml/min (according to the CKD-EPI formula)

Exclusion criteria:

* Known allergies or intolerance to one or more compounds present in one of the first line or second line regimens
* Concomitant need for full anticoagulation that cannot be interrupted or bridged prior to tissue biopsy
* ECOG PS >2
* Heart failure (NYHA class III-IV)
* Severe or uncontrolled concurrent illness
* Active viral infection from HIV, HBV or HCV, even if under antiretroviral treatment
* Myocardial infarction within the previous 6 months
* Patients who are pregnant or breastfeeding

ELIGIBILITY:
Inclusion criteria:

* Informed Consent as documented by signature
* Patients older than 18 years
* Patients with metastatic pancreatic ductal adenocarcinoma
* At least one lesion amenable for surgical excisional biopsy
* ECOG Performance status 0-2
* Radiologically measurable disease
* Life expectancy > 3 months
* Absolute leucocyte count >1.5 G/l, platelets >100 G/l
* Serum creatinine <1.5 times of the upper limit of normal or Clearance >50ml/min (according to the CKD-EPI formula)

Exclusion criteria:

* Known allergies or intolerance to one or more compounds present in one of the first line or second line regimens
* Concomitant need for full anticoagulation that cannot be interrupted or bridged prior to tissue biopsy
* ECOG PS >2
* Heart failure (NYHA class III-IV)
* Severe or uncontrolled concurrent illness
* Active viral infection from HIV, HBV or HCV, even if under antiretroviral treatment
* Myocardial infarction within the previous 6 months
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with the diagnosis of metastatic adenocarcinoma of the pancreas can be enrolled provided the above mentioned criteria apply.
  The patients can either be therapy-naive or pretreated.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Is there a significant correlation between Oncotarget/Oncotreat based predicted drug sensitivity and the patient's progression-free survival (PFS) in metastatic pancreatic adenocarcinoma after administered standard therapy ? | From enrollment to disease progression according to the RECIST v1.1 criteria, assessed up to 100 months
  To demonstrate a significant correlation between the degree of sensitivity predicted by Oncotreat/Oncotarget to Gemcitabine-Abraxane, or Abraxane-Gemcitabine-FOLFOX (according to the SEQUENCE trial) or FOLFIRINOX (according to the NAPOLI-3 trial), and clinical progression free survival (PFS) in metastatic pancreatic adenocarcinoma.

SECONDARY OUTCOMES:
1) Correlation between Darwin-test predicted drug sensitivity and patient-derived PDO sensitivity to clinically used drug regimens. 2) Correlation between the measured PDO sensitivity to the administered standard therapies 3) Biobanking | Observation until progression under given standard treatment using RECIST and TU markers. Follow up until progression and/or death at least 60 months.
  We will analyze if Darwin and PDO prediction are similar or different with regard to the observed chemrsensitivity under a given standard regimen.
  We will then also analyze if PDO prediction is reflected in the clinical course of the patient. Tissue and blood samples are stored for Biobanking.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Schmidt, Prof. Dr. med. Dres. h.c., MME, Study Director — Swiss Surgery/Hirslanden Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Morikawa T, Yoshida M. A useful testing strategy in phase III trials: combined test of superiority and test of equivalence. J Biopharm Stat. 1995 Nov;5(3):297-306. doi: 10.1080/10543409508835115. PMID 8580930
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Paluri RK, Kasi A, Young C, Posey JA. Second-line treatment for metastatic pancreatic cancer. Clin Adv Hematol Oncol. 2020 Feb;18(2):106-115. PMID 32558804
- [Result] Ettrich TJ, Seufferlein T. Systemic Therapy for Metastatic Pancreatic Cancer. Curr Treat Options Oncol. 2021 Oct 19;22(11):106. doi: 10.1007/s11864-021-00895-4. PMID 34665339
- [Result] Zhang XW, Ma YX, Sun Y, Cao YB, Li Q, Xu CA. Gemcitabine in Combination with a Second Cytotoxic Agent in the First-Line Treatment of Locally Advanced or Metastatic Pancreatic Cancer: a Systematic Review and Meta-Analysis. Target Oncol. 2017 Jun;12(3):309-321. doi: 10.1007/s11523-017-0486-5. PMID 28353074
- [Result] Nguyen KT, Gamblin TC, Geller DA. World review of laparoscopic liver resection-2,804 patients. Ann Surg. 2009 Nov;250(5):831-41. doi: 10.1097/SLA.0b013e3181b0c4df. PMID 19801936
- [Result] Strassburg CP, Manns MP. Approaches to liver biopsy techniques--revisited. Semin Liver Dis. 2006 Nov;26(4):318-27. doi: 10.1055/s-2006-951599. PMID 17051446
- [Result] Vasciaveo A, Arriaga JM, de Almeida FN, Zou M, Douglass EF, Picech F, Shibata M, Rodriguez-Calero A, de Brot S, Mitrofanova A, Chua CW, Karan C, Realubit R, Pampou S, Kim JY, Afari SN, Mukhammadov T, Zanella L, Corey E, Alvarez MJ, Rubin MA, Shen MM, Califano A, Abate-Shen C. OncoLoop: A Network-Based Precision Cancer Medicine Framework. Cancer Discov. 2023 Feb 6;13(2):386-409. doi: 10.1158/2159-8290.CD-22-0342. PMID 36374194
- [Result] Yang H, Sun L, Liu M, Mao Y. Patient-derived organoids: a promising model for personalized cancer treatment. Gastroenterol Rep (Oxf). 2018 Nov;6(4):243-245. doi: 10.1093/gastro/goy040. Epub 2018 Oct 9. No abstract available. PMID 30430011
- [Result] Tiriac H, Bucobo JC, Tzimas D, Grewel S, Lacomb JF, Rowehl LM, Nagula S, Wu M, Kim J, Sasson A, Vignesh S, Martello L, Munoz-Sagastibelza M, Somma J, Tuveson DA, Li E, Buscaglia JM. Successful creation of pancreatic cancer organoids by means of EUS-guided fine-needle biopsy sampling for personalized cancer treatment. Gastrointest Endosc. 2018 Jun;87(6):1474-1480. doi: 10.1016/j.gie.2017.12.032. Epub 2018 Jan 9. PMID 29325707
- [Result] Rawla P, Sunkara T, Gaduputi V. Epidemiology of Pancreatic Cancer: Global Trends, Etiology and Risk Factors. World J Oncol. 2019 Feb;10(1):10-27. doi: 10.14740/wjon1166. Epub 2019 Feb 26. PMID 30834048
- [Result] Ilic M, Ilic I. Epidemiology of pancreatic cancer. World J Gastroenterol. 2016 Nov 28;22(44):9694-9705. doi: 10.3748/wjg.v22.i44.9694. PMID 27956793
- [Result] Emanuel EJ, Wendler D, Grady C. What makes clinical research ethical? JAMA. 2000 May 24-31;283(20):2701-11. doi: 10.1001/jama.283.20.2701. PMID 10819955